CLINICAL TRIAL: NCT00707408
Title: A Phase II Trial Evaluating the Safety and the Efficacy of High-Dose Imatinib in Relapsed/Refractory c-Kit Positive and BCR-Abl Negative AML Patients
Brief Title: High-Dose Imatinib for Relapsed/Refractory c-Kit Positive Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Dr Patrice Chevallier
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 03/3-B
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: AML
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Imatinib — Daily dosing of imatinib 600 mg/day is planned for one month or until progression of disease. Dose increase to 800 mg/ day imatinib is permitted for 2 additional months in the event of response failure. Novartis provided supplies of imatinib for all patients included in the study.

SUMMARY:
This is a multicenter open-label phase II trial of high dose imatinib mesylate in patients with AML in first or second relapse, or with refractory disease. Daily dosing of imatinib 600 mg/day is planned for one month or until progression of disease. Dose increase to 800 mg/ day imatinib is permitted for 2 additional months in the event of response failure. Response is assessed after 1, 2 and 3 months of treatment by bone marrow aspirate.

DETAILED DESCRIPTION:
Daily dosing of imatinib 600 mg/day is planned for one month or until progression of disease. Dose increase to 800 mg/ day imatinib is permitted for 2 additional months in the event of response failure. Novartis provided supplies of imatinib for all patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* AML in first or second relapse,
* refractory AML
* performance status of 0-2 on the Eastern Cooperative Oncology Group scale,
* adequate hepatic and renal functions (AST or ALT <= 5 times the upper limit of normal
* creatinine < 2 times the upper limit of normal)

  * 20% blasts in bone marrow,
  * 70% of bone marrow blast population c-kit positive as assessed by immunophenotyping
* Bcr-Abl negative chromosomal analysis (assessed by fluorescence in situ hybridization; FISH), and no chromosome 5-12 translocation

Exclusion Criteria:

* Previous treatment by Imatinib
* Secondary AML

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-02; Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hopspital, Nantes, France